CLINICAL TRIAL: NCT01373645
Title: Safety and Efficacy Registry of Yinyi Polymer-free Paclitaxel-eluting Stent
Brief Title: Safety and Efficacy Registry of Yinyi Stent
Acronym: SERY-I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Weifeng Shen, Ruijin hospital, shanghai jiao tong university school of medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH20100909
Record Dates: First submitted 2011-04-01; First posted 2011-06-15 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (1):
- Yinyi stent (Experimental): subjects with Yinyi stent implantation
  Interventions: Device: Yinyi stent

INTERVENTIONS:
Device: Yinyi stent — subjects with Yinyi stent implantation

SUMMARY:
Drug-eluting stents effectively reduce restenosis but may increase late thrombosis and delayed restenosis. Persistent polymer could be responsible. Local delivery of paclitxel from a polymer-free Yinyi stent (Dalian Yinyi biomaterial research and development co.ltd) may prevent these complications.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old
* both gender
* native coronary lesion
* narrowing > 70%
* vessel size 2.5-4.0 in diameter

Exclusion Criteria:

* without informed consent,
* ST elevation myocardial infarction within 7 days,
* patient with ≤ 70% coronary narrowing at target lesion,
* left main lesion,
* multivessel narrowing need more than 3 stent implantations,
* by-pass graft,
* abnormal liver function before randomization,
* active hepatitis or muscular disease,
* impaired renal function with serum creatinine level > 3mg/dl,
* impaired left ventricular function with LVEF < 30%,
* Participate in other studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac events | 12 months
  including cardiac death, myocardial infarction and target vessel failure

SECONDARY OUTCOMES:
stent thrombosis | 12 months
  according to ARC definition

CONTACTS AND LOCATIONS:
Locations (1):
- ruijin hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Zhang RY, Zhang Q, Zhu JZ, Chen LL, Zhang CY, Zhou XC, Yuan Y, Zhong ZX, Li L, Qiu J, Wang W, Chen XM, Yang ZJ, Yan JC, Chen SL, Hou YQ, Wu YQ, Luo HM, Qiu JP, Zhu L, Wang Y, Fu GS, Wang JA, Ma KH, Yin YH, Zhang DF, Hu XS, Zhu GY, Shen WF; Safety and Efficacy Registry of Yinyi stent (SERY-I) Investigators. Safety and efficacy of polymer-free paclitaxel-eluting microporous stent in real-world practice: 1-year follow-up of the SERY-I registry. Chin Med J (Engl). 2011 Nov;124(21):3521-6. No abstract available. PMID 22340171